CLINICAL TRIAL: NCT05981352
Title: Clinical, Radiographic and Microbiological Evaluation of Hyaluronic Acid and Amniotic Membrane Allograft in Comparison to Mineral Trioxide Aggregate in Pulpotomy of Primary Molars (Randomized Clinical Trial and In Vitro Study)
Brief Title: Evaluation of Different Materials in Pulpotomy of Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pulpotomy of Primary Molars
Record Dates: First submitted 2023-01-26; First posted 2023-08-08 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-05

CONDITIONS: Pulp Disease, Dental
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Mineral trioxide aggregate (positive control group) (Active Comparator): : according to the manufacturing instructions as following:
  * After achieving hemostasis, Mineral trioxide aggregate powder will be mixed with saline.
  * Then Mineral trioxide aggregate will be placed directly on the pulp stumps.
  Interventions: Procedure: mineral trioxide aggregate pulpotomy
- Dehydrated amniotic membrane group (Experimental): * After achieving hemostasis, a double layer of sterile processed human allograft tissue (dehydrated dual-layer dental amnion patch) will be trimmed and soaked in saline for a minute.
  * Dehydrated amniotic membrane will be Placed directly on the pup stumps using sterile tweezers and adjusted to the entire floor of the pulp chamber.
  Interventions: Procedure: Dehydrated amniotic membrane pulpotomy
- Hyaluronic acid group (Experimental): • After achieving hemostasis, pulp stumps will be covered with a mixture of Hyaluronic acid gel and zinc oxide powder with consistency (1:1 ratio by volume) .
  Interventions: Procedure: Hyaluronic acid pulpotomy

INTERVENTIONS:
Procedure: mineral trioxide aggregate pulpotomy — * After achieving hemostats, Mineral trioxide aggregate powder will be mixed with saline.
  * Then Mineral trioxide aggregate will be placed directly on the pulp stumps.
  Arms: Mineral trioxide aggregate (positive control group)
Procedure: Dehydrated amniotic membrane pulpotomy — * After achieving haemostasis, a double layer of sterile processed human allograft tis¬sue (dehydrated dual-layer dental amni¬on patch) will be trimed and soaked in saline for a minute.
  * Dehydrated amniotic membrane will be Placed directly on the pup stumps using sterile tweezers and adjust¬ed to the entire floor of the pulp chamber.
  Arms: Dehydrated amniotic membrane group
Procedure: Hyaluronic acid pulpotomy — * After achieving haemostasis, pulp stumps will be covered with a mixture of Hyaluronic acid gel and zinc oxide powder with consistency (1:1 ratio by volume) .
  * The cavities of all pulpotomy molars will be sealed with a layer of reinforced zinc oxide and eugenol .
  Arms: Hyaluronic acid group

SUMMARY:
The aim of the current study is to evaluate and compare clinical and radiographic success and antibacterial effect of Hyaluronic Acid and Amniotic membrane pulpotomy in primary molars in comparison with MTA pulpotomy (Randomized Clinical Trial and In Vitro Study).

DETAILED DESCRIPTION:
Pulpotomy is one of the most used frequently treatment for pulp involved in primary teeth. Pulpotomy is performed in a primary tooth with extensive caries but without evidence of radicular pathology when caries removal results in a carious or mechanical pulp exposure. It is a conservative therapy performed to remove the inflamed coronal pulp tissues followed by application of an effective and compatible bactericidal medicament.

Many different compounds have been suggested include glutaraldehyde, electrosurgery, calcium hydroxide, ferric sulfate, freeze-dried bone, bone morphogenic proteins (BMP), mineral trioxide aggregate (MTA) and Bio dentine (Tricalcium Silicate Cement) as replacement for Form cresol in pulpotomy procedure however.

Pulpotomy has been broadly classified as devitalization, preservation, and regeneration of the remaining pulp tissue. Other materials that has shown immense potential for regeneration like mineral trioxide aggregate (MTA). It is a biocompatible and bio inductive material that has been investigated for endodontic.

Hyaluronic acid (HA) has recently emerged as a material of choice in preserving the vitality of the pulp. It is a natural mucopolysaccharide, carbohydrate polymer from the group of glycosaminoglycans. HA is synthetized on the cytoplasmic surface of plasma membranes and is common in humans and other vertebrates. It is the major component of the inner-cell cement of the capillary wall, and of the extracellular matrix of the connective tissue. Deposition of HA significantly increases during development, morphogenesis, wound repair and regeneration, malignancy, and inflammation.

Hyaluronic acid (HA) or hyaluronan is a hydrated anionic polysaccharide plentiful in the extracellular matrix with a molecular weight of 4000-20,000,000 Da that is found in a variety of tissues including skin, synovial fluid, cartilage, tendons, eyes and embryonic mesenchyme . It is comprised of repeating disaccharides d-glucuronic acid and N-acetyl-d-glucosamine, which are joined together by alternating β-1,4 and β-1,3 glycoside bonding. During bone repair, it encourages the undifferentiated mesenchymal cells to migrate, adhere, and proliferate into osteoblastic cells. Due to its non-toxicity, biocompatibility, biodegradability and non-immunogenicity, and used in ophthalmology and orthopedics as an anti-inflammatory agent and anti bacterial agent.

The use of a hyaluronic acid to cover a dentin defect, stimulated a cell-rich rearrangement of pulp tissue with few inflammatory cells, as well as being an acceptable and biocompatible scaffold for regenerating the dental pulp. Because of its high molecular weight when dissolved in water, hyaluronic acid's viscoelasticity increases, making it simpler to use as an injectable scaffold. Moreover, advantageous characteristics are related to the hyaluronic acid scaffolds as bioactivity, biocompatibility, biodegradability, in addition to serving as a reservoir for growth factors..

It is important to propose new biologically based therapeutics directed at preserving pulp vitality , forming biological tissue and neutralizing the side effects of previously used synthetically based biomaterials .

Recently, novel biologically based materials have been developed from the placenta or other gestational tissues like the umbilical cord with highly rich stem cell reservoirs . Amniotic membrane (AM) is a fetes membranous sac forming the innermost layer of the placenta. It is a bi-layered membrane consists of amnion and chorion. Amnion consists of 3 distinct thin layers: an epithelial monolayer (closest to the fetes),a basement membrane and avascular mesenchymal stromal matrix (containing mesenchymal stem cells) that composed of 3 adjacent but distinct layers: outermost spongy, middle fibroblastic and inner compact.

Although it is a thin membrane (70-180 μm thick), it is remarkably elastic and strong natural biological barricade protecting the fetus from trauma and bacterial infection . In contrast, the chorion is 3-4 times thicker than amnion and consists of a reticular, basement membrane, and trophoblastic layers. Both membranes play important roles in embryo's overall development, embryo's nourishment and breathing .

Amniotic membrane matrix contains plenteous growth factors (GFs) including basic-fibroblast growth factor (b-FGF), nidogen growth factor (NGF), keratinocyte growth factor (KGF), epidermal derived growth factor (EDGF), and transforming GF-beta growth factor (TGF-β) which promote tissue regeneration . These GFs mimic the stem cell niche for ex vivo growth and provide a natural healing environment. It acts as a structural scaffold supporting proliferation, differentiation, and regeneration due to presence of fibronectin, laminins, proteoglycans, collagen types I, III, IV, V and VI, elastin, nidogen, and hyaluronic acid in its stromal layer, and act as an excellent candidature for a native scaffold in tissue engineering .

Furthermore, it secretes nutrient factors , promotes cell migration, adhesion, differentiation, and suppresses the semi allogenic immune response against the foetus . In addition, it has a biological, anti-inflammatory (similar to cortisone and steroids shots), anti-fibrotic, anti-microbial (including beta-defensins), anti-scarring, anti-angiogenic and analgesic properties that make it a unique therapy for wound care and ideal substrate for supporting the growth of mesenchymal progenitor cells via prolonging their lifespan

It is used in allotransplant due to its ability to promote cellular growth and attachment with the lack of its immunogenicity and toxicity; it was first reported by Davis since 1910 in skin transplantation. Also, it has been used successfully for over a decade in a wide range of surgical application, biological wound dressing, ophthalmic reconstructive surgery, an adhesion barrier in the spine, and in-ear and orthopedic surgery. It is easily obtained, processed, transported, and prepared in different forms for clinical use like fresh, dried, frozen, freeze derived irradiated, stabilized amniotic and cryopreserved membranes .

Amnion-based products have a proven rate of success in the field of dentistry since 1990s, when first demonstrated safety and efficacy in pre-and clinical studies . The dehydrated or cryopreserved membrane is used for retaining the majority of the natural (fibrillar and membranous) collagens, maintaining the composition of GFs and bioactive molecules found in natural and unprocessed placental tissues, and increasing stability and shelf life of the product .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 4 to 8 years old.
* Patients who are free from ant medical condition.
* Patients who have a vital deep carious Mandibular primary molar which is indicated for pulpotomy .
* No clinical signs or symptoms of irreversible pulpitis as pain on percussion, tooth mobility, presence of sinus or fistula, history of swelling , Spontaneous pain.
* No radiographic evidence of any periapical pathosis , Internal or external root resorption , Absence of discontinuity of lamina dura .
* Physiological root resorption not more than 1/3 of crown

Exclusion Criteria:

* Teeth that are badly broken down, that cannot be restored.
* Presence of uncontrolled bleeding after pulpotomy
* Patients/ parent guardians that refuse to sign informed consent.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
clinical pulp testing | 0 baseline , changes from baseline pulp condition at 3 month, change from the baseline pulp condition at 6 month, change from baseline pulp condition at 9 month, change from base line pulp condition at 12 month.
  pulp testing clinically measured by zurn and seale criteria ,
Radio graphic pulp testing | 0 baseline , changes from baseline pulp condition at 3 month, change from the baseline pulp condition at 6 month, change from baseline pulp condition at 9 month, change from base line pulp condition at 12 month.
  pulp testing radio graphic measured by digital radio graph parallel technique

CONTACTS AND LOCATIONS:
Overall Officials: eman Ib Abdel Maksoud, doctor, Study Chair — Ain Shams University